CLINICAL TRIAL: NCT01024296
Title: Pivotal Study to Evaluate the Efficacy of a Laparoscopic Port Closure Device
Brief Title: Efficacy Study to Evaluate Laparoscopic Fascial Closure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: SurgSolutions, LLC (Industry)
Responsible Party: Principal Investigator, Thomas Krummel, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-11062009-4361; IRB Protocol #8864 (Other: Stanford University)
Record Dates: First submitted 2009-11-13; First posted 2009-12-02 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Hernia, Abdominal
MeSH Terms: conditions — Hernia, Abdominal

ARMS (1):
- Gastric Bypass Surgery Patients (Experimental): Surgical site closure using Port Close device
  Interventions: Device: Port Close

INTERVENTIONS:
Device: Port Close — Device for applying loop suture to close surgical site

SUMMARY:
During any minimally invasive surgery case, 5-25mm size incisions need to be made to gain access to the abdomen. One of the most difficult, time-consuming, and sometimes unreliable parts of the case is closing these incisions, especially in obese patients. This is mainly because these incisions are very small and the layer that needs to be closed (fascia) rests deep underneath the skin and fat tissue of the abdominal wall. Two of the investigators (CM and BS) have developed at Stanford an instrument that allows for an easier and more reliable closure of these wounds. The purpose of this study is to test this instrument in the closure of laparoscopic wounds in obese patients undergoing laparoscopic gastric bypass surgery.

DETAILED DESCRIPTION:
For the patients enrolling in this study, preoperative and postoperative care will be exactly the same. The operative procedure will also be very similar with the only modification being in the way the ports are closed at the end of the surgery and the fact that all ports 11mm or greater will be closed (instead of leaving 11 or 12mm ports to be closed at the discretion of the surgeon). Instead of using a suture-passer to place the suture through the fascia, the surgeon will use the new instrument to drive the suture into the tissue under direct visualization through the umbilical port camera. The same instrument but with new sutures will be used for each of the interrupted stitches that are usually placed to close the port.

The instrument that has been developed by some of the investigators is a 10mm elongated device that can easily be inserted into the port or fascial opening. If inserted through the port, the trocar can then be slid over the instrument to remove the trocar without losing pneumoperitoneum. The instrument has two opposing wings that will open once placed beyond the fascial opening. As the surgeon pulls up on the device, the wings open sliding along the fascia and pushing away any intra-abdominal contents that may be close to the instrument. Once the surgeon assures under direct visualization with the camera that the wings are open at both sides of the wound and that all intra-abdominal contents are out of the way (just as the surgeon would with the standard technique), he or she pushes a plunger that drives two flexible nitinol needles from the shaft of the instrument, through the fascia, and into the wings. The needles will be received in the wings by a set of couplers attached to the same suture that would be used otherwise (#0 Vycril). The surgeon then releases the wings and pulls out the device, leaving a looped suture placed around the opening. The surgeon can then tie the sutures as he or she would normally do on the standard procedure. At any time, the surgeon can reposition or remove the instrument without placing the sutures. The procedure may be repeated as many times as the surgeon considers necessary (usually 1 to close the 11 or 12mm fascial ports and 2 or 3 to close the 25mm fascial port).

ELIGIBILITY:
Inclusion Criteria:- Clinical Diagnosis of Morbid Obesity

* BMI > 40 or BMI > 35 with medical comorbidities
* Undergoing laparoscopic gastric surgery
* Have at least one trocar site measuring 12 mm or greater Exclusion Criteria:Vulnerable subjects will be excluded including:

  1. Children
  2. Pregnant women
  3. Economically and educationally disadvantaged
  4. Decisionally impaired
  5. Homeless people
  6. Employees and students.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Krummel, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gastric Bypass Surgery Patients
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Successful Port Site Closure Using Port Close Device
Time Frame: Day 1, at the end of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 4
Participants | 3

2. Primary Outcome: Time of Port Site Closure
Time Frame: Day 1, from insertion to removal of Port Close device during surgery
Population: Participants with successful closure using the Port Close device were included in the analysis.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 3
seconds | 138.7 (22.21)

ADVERSE EVENTS:
Arm/Group | Gastric Bypass Surgery Patients
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes